CLINICAL TRIAL: NCT04133896
Title: Circulating IL-6, Clusterin and Irisin in Obese Subjects With Different Grades of Obesity: Association With Insulin Resistance and Sexual Dimorphism
Brief Title: Circulating IL-6, Clusterin and Irisin in Obese Subjects
Status: Completed | Type: Observational
Sponsor: Rehab Werida (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Clinical Pharmacy Lecturer, Damanhour University
Organization: Damanhour University (Other)
Other Study IDs: Obesity and IR
Record Dates: First submitted 2019-10-18; First posted 2019-10-21 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Group 1 Male: group 1 (22 lean men),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 2 Male: group 2 (22 class I obese men),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 3 Male: group 3 (22class II obese men),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 4 Male: group 4 (22 class III obese men).
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 1 Female: group 1 (22 lean women),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 2 Female: group 2 (22 class I obese women),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 3 Female: group 3 (22 class II obese women),
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level
- Group 4 Female: group 4 (22 class III obese women).
  Interventions: Diagnostic Test: IL-6, Clusterin, Irisin Level

INTERVENTIONS:
Diagnostic Test: IL-6, Clusterin, Irisin Level — Blood samples to determine levels of Circulating IL-6, Clusterin and Irisin

SUMMARY:
evaluate the circulating levels of IL-6, clusterin and irisin in obese subjects of both sexes who had different classes of obesity and their sexual dimorphism also identify the association of IL-6, clusterin and irisin with insulin resistance.

DETAILED DESCRIPTION:
Aim: Firstly, this study aimed at assessing the circulating levels of IL-6, clusterin and irisin in obese subjects of both sexes who had different classes of obesity and evaluating their sexual dimorphism and secondly evaluate the association of IL-6, clusterin and irisin with insulin resistance.

Method: This study was conducted on 176 non-diabetic subjects of both sexes. Participants were classified according to their sex into two groups; the male and female groups. The male group (88 men) was classified according to BMI into; group 1 (22 lean men), group 2 (22 class I obese men), group 3 (22 class II obese men), and group 4 (22 class III obese men). The female group (88 women) was also classified according to BMI exactly as the male group. Fasting blood glucose, fasting insulin, lipid panel, serum IL-6, clusterin and irisin levels were measured. One-way analysis of variance followed by Tukey's as post hoc test was used for comparison of variables.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Female and Male
* Age matched adult non-diabetic non-smoker males and females'

Exclusion Criteria:

* smokers, subjects with a history of diabetes mellitus, liver, renal, thyroid, inflammatory diseases, and females on contraceptives pills. Patients on medications that can interfere with glucose or lipid metabolism (corticosteroids, anti-hyperlipidemics, non-selective beta blockers, thiazides, etc.) and subjects with organic causes of obesity were also excluded from this study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — based on self-representation of gender identity.
Study Population: Subjects included in the study were classified according to their sex into two main group the male group and the female group. The male group contained 88 men which subdivided according to the BMI into the following groups; group 1 (22 lean men), group 2 (22 class I obese men), group 3 (22class II obese men), and group 4 (22 class III obese men). The female group contained 88 adult women which sub-classified according to BMI into the following subgroups; group 1 (22 lean women), group 2 (22 class I obese women), group 3 (22 class II obese women), and group 4 (22 class III obese women).
Sampling Method: Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
insulin resistance | 18 months
  by homeostasis insulin resistance index (fasting insulin (μIU/ml) times fasting glucose (mg/L) divided by 405 )
IL- 6 | 18 Months
  blood level of IL-6
Clusterin | 18 Months
  blood level of Clusterin
Irisin | 18 Months
  blood level of Irisin
Lipid profile | 18 Months
  Plasma triglycerides and total cholesterol were measured by enzymatic colorimetric method. High-density lipoprotein cholesterol (HDL-C) was measured by precipitation method. Low density lipoprotein cholesterol (LDL-C) was calculated using the Friedewald formula

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Lecturer, Principal Investigator — Damanhour University, Faculty of Pharmacy
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gouni-Berthold I, Berthold HK, Huh JY, Berman R, Spenrath N, Krone W, Mantzoros CS. Effects of lipid-lowering drugs on irisin in human subjects in vivo and in human skeletal muscle cells ex vivo. PLoS One. 2013 Sep 2;8(9):e72858. doi: 10.1371/journal.pone.0072858. eCollection 2013. PMID 24023786
- [Result] Baralla A, Sotgiu E, Deiana M, Pasella S, Pinna S, Mannu A, Canu E, Sotgiu G, Ganau A, Zinellu A, Sotgia S, Carru C, Deiana L. Plasma Clusterin and Lipid Profile: A Link with Aging and Cardiovascular Diseases in a Population with a Consistent Number of Centenarians. PLoS One. 2015 Jun 15;10(6):e0128029. doi: 10.1371/journal.pone.0128029. eCollection 2015. PMID 26076476
- [Result] van Greevenbroek MM, Schalkwijk CG, Stehouwer CD. Obesity-associated low-grade inflammation in type 2 diabetes mellitus: causes and consequences. Neth J Med. 2013 May;71(4):174-87. PMID 23723111